CLINICAL TRIAL: NCT04533152
Title: Prognostic Determinants in Patients With Diabetic Foot Ulcer (PDF Cohort) - A French Prospective Multicentre Cohort.
Brief Title: Prognostic Determinants in Patients With Diabetic Foot Ulcer.
Acronym: PDF
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Fondation Francophone pour la Recherche sur le Diabete (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2019/70
Record Dates: First submitted 2020-08-27; First posted 2020-08-31 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Diabetic Foot Ulcer
Keywords: Diabetes mellitus; Lower-limb amputation; Wound; Health-related quality of life; Cost-of-illness
MeSH Terms: conditions — Diabetic Foot; Diabetes Mellitus; Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 1 PAXgene blood DNA tube (2.5 mL)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The worse prognosis observed in patients with Diabetic Foot Ulcer (DFU) has not been fully understood. Poor prognosis may be related to other conditions (inflammation, infectious disease, cancers) further to cardiovascular disease.

The aim of the study is to conduct the first prospective, observational and multi-centre cohort of patients with DFU in France, in order to evaluate the 5-years mortality rate, its causes and relevant prognostic determinants.

DETAILED DESCRIPTION:
Diabetic foot ulcer (DFU) is one of the major complications frequently observed in patients with diabetes. DFU is the leading cause of non-traumatic lower-limb amputation (LLA), and it is associated with cognitive decline, worsening quality of life and substantial economic impact on French healthcare system. DFU is also associated with excess risk of premature death with significant decrease in life expectancy despite major improvement in medical care during last decades. The hypothesis of the study is that this worse prognosis seen in DFU patients may not be fully explained by a high cardiovascular risk, but mainly linked to different causes, including inflammatory, infectious and malignant conditions.

In addition, to conduct the first prospective, observational and multi-centre cohort of patients with DFU in France to evaluate the 5-years mortality rate, its causes and relevant prognostic determinants, the investigators will also assess all changes in health-related quality of life (HRQoL), and the economic impact related to DFU (cost of illness study) for the French healthcare system, using SNDS claims databases. A 3-year inclusion period will start during 2020, and each participant will be followed for 5 years or until death.

ELIGIBILITY:
Inclusion Criteria:

Adults with diabetes and DFU, defined as a foot skin ulceration or open LLA wound, measuring at least 5 mm of diameter, located below the malleolus, and induced by diabetic complications. In the case of an amputation before inclusion, the amputation stump will be considered as the main wound and not the wound that led to the amputation.

Exclusion Criteria:

* Acute or chronic lower-limb ischemia without open skin wound,
* Foot infection without open skin wound,
* Intercurrent disease prohibiting participation in an observational study,
* Pregnancy or breastfeeding
* Curatorship or guardianship
* Prisoners -- Patient currently participating to more than one other clinical study (interventional or observational, 2 study maximum including PDF) or currently participating to another study interfering with standard care of diabetic foot

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: PDF study is designed to be the first French multicentre, observational and prospective cohort of patients with DFU referred from the community into secondary and tertiary care foot clinics.
  Twenty-three French centres agreed to participate in this study. Each centre will recruit during the 3-year inclusion period.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-11-24 (Actual); Primary Completion 2029-11 (Estimated); Study Completion 2029-11 (Estimated)

PRIMARY OUTCOMES:
DFU risk score | 5 years after inclusion
  Construct a DFU risk score equation of all-death will be computed to determine individuals with the higher risk of worse outcomes.

SECONDARY OUTCOMES:
Survival without active index DFU | At 3 and 12 months after inclusion day
Survival without recurrent index DFU | At 12, 24, 36, 48, 60 months after inclusion day
Survival without major adverse limb events (MALE) | 5 years after inclusion
  MALE is a composite of foot infection, non-traumatic lower-limb amputation (LLA), requirement of revascularization, whichever comes first. These components will be also considered individually.
Survival without major macrovascular events (MACE) | 5 years after inclusion
  MACE is a composite of non-fatal myocardial infarction, non-fatal stroke, hospitalization for heart failure, or cardiovascular death, whichever comes first.
Survival without major microvascular events (MICE) | 5 years after inclusion
  MICE is a composite of new-onset persistent macroalbuminuria, sustained 40% declined eGFR from baseline, ESRD, severe diabetic retinopathy or macular oedema requiring laser photocoagulation or intravitreal therapies, or diabetes-related blindness in either eye, whichever comes first.

CONTACTS AND LOCATIONS:
Locations (26):
- France (25):
  - CHU Côte de Nacre, Caen
  - CH Sud Francilien, Corbeil-Essonnes
  - CHU de Bocage Sud, Dijon
  - CHU de La Réunion - Site Sud, La Réunion
  - Groupe Hospitalier de La Rochelle Ré Aunis, La Rochelle
  - Hôtel Dieu, Le Creusot
  - CHRU de Lille - Hôpital Claude Huriez, Lille
  - AP - HM - Hôpital de la Conception, Marseille
  - CHU de Montpellier - Hôpital Lapeyronie, Montpellier
  - CHU de Nantes Hôpital Nord Laennec, Nantes
  - CH Pierre Bérégovoy, Nevers
  - CHU de Nice - Hôpital l'Archet 2, Nice
  - CHU Nîmes - Hôpital universitaire Carémeau, Nîmes
  - AP-HP - Hôpital Bichat, Paris
  - AP-HP - Hôpital Lariboisière, Paris
  - AP-HP - Hôpital Pitié-Salpétrière, Paris
  - Hôpital Paris Saint Joseph, Paris
  - Hopital Haut-Leveque, Pessac
  - HCL - Hôpital Lyon sud, Pierre-Bénite
  - CHU de la Milétrie, Poitiers
  - CHU de Rouen, Rouen
  - Centre Hospitalier Saint Benoit, Saint-Benoît
  - Hôpital d'Instruction des Armées Bégin, Saint-Mandé
  - Maison de Santé Protestante Bagatelle - Hôpital Bagatelle, Talence
  - CHU de Toulouse - Hôpital Rangueil, Toulouse
- CHU de la Martinique, Fort-de-France, Martinique